CLINICAL TRIAL: NCT05124509
Title: Immune Response to Third Dose of SARS-CoV-2 Vaccine in a Cohort of Solid Organ Transplant Recipients
Brief Title: Immune Response to Third Dose of COVID-19 Vaccine in Solid Organ Transplant
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 210405014E
Record Dates: First submitted 2021-11-15; First posted 2021-11-18 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; SARS-CoV-2 Infection; Solid Organ Transplant; Vaccine Response Impaired
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Three doses of BNT162b2 vaccine: Solid organ transplant patients who received three doses of BNT162b2
  Interventions: Biological: Three doses of SARS-CoV-2 BNT162b2 vaccine (observational)
- Two doses of Coronavac and one of BNT162b2 vaccine: Solid organ transplant patients who received two doses of CoronaVac and one dose of BNT162b2
  Interventions: Biological: Two doses of CoronaVac and one dose of BNT162b2 SARS-CoV-2 vaccine (observational)

INTERVENTIONS:
Biological: Three doses of SARS-CoV-2 BNT162b2 vaccine (observational) — Two doses of SARS-CoV-2 BNT162b2 mRNA vaccine, followed by a booster (3rd) dose of SARS-CoV-2 BNT162b2 mRNA vaccine.
  Groups: Three doses of BNT162b2 vaccine
Biological: Two doses of CoronaVac and one dose of BNT162b2 SARS-CoV-2 vaccine (observational) — Two doses of CoronaVac SARS-CoV-2 inactivated vaccine, followed by a booster (3rd) dose of BNT162b2 mRNA vaccine.
  Groups: Two doses of Coronavac and one of BNT162b2 vaccine

SUMMARY:
The Coronavirus Disease 2019 (COVID-19) pandemic has claimed over 5 million lives globally. Fortunately, a substantial and growing number of SARS-CoV-2 vaccines with very high efficacy have been developed, manufactured, and rapidly approved. Novel mRNA vaccines such as the BNT162b2 (Pfizer-BioNTech) and mRNA-1273 (Moderna) have reported a stunning >94% efficacy against COVID-19. However, global access has not been equitable, with many low- and middle-income countries having no vaccine access or access under emergency use mainly to traditional inactivated SARS-CoV2-2 vaccines such as BBIBP-CorV (Sinopharm Beijing), CoronaVac (Sinovac) and BBV152 (Bharat Biotech). Emerging studies have shown that lower concentrations of neutralizing antibodies (Nab) are attained after CoronaVac than after an mRNA-based vaccine in healthy individuals. This difference seems to be more pronounced in immunocompromised patients who are at higher risk of severe COVID-19 and death from COVID-19. As such, several countries including the United States, Israel and Chile have recommended a third vaccine dose for high-risk populations. However, it is not currently known which is the best vaccine combination regarding immunogenicity, particularly in these vulnerable patients.

This observational study will explore the humoral and cellular response to a SARS-CoV-2 BNT162b2 vaccine booster in solid organ transplant patients who received two previous doses of the inactivated Coronavac or two doses of BNT162b2 vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Solid organ transplant patients in the last 10 years and currently under immunosuppressive therapy
* Vaccination with two doses of Coronavac vaccine or BNT162b2 vaccines, followed by a booster dose (3d dose) of BNT162b2 vaccine administered in the previous 8-12 weeks.

Exclusion Criteria:

* Previous SARS-CoV-2 infection
* Booster vaccine (3rd dose) administered less than 8 weeks or more than 12 weeks before enrolment
* Intravenous immunoglobulin therapy 60 days before enrolment
* Previous SARS-CoV-2 vaccine different from CoronaVac or BNT162b2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Solid organ transplant patients in the last 10 years and currently under immunosuppressive therapy
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
IgG seropositivity 8-12 weeks after third dose BNT162b2 (booster) vaccine. | 8-12 weeks after booster vaccine

SECONDARY OUTCOMES:
Proportion of positive neutralizing antibodies 8 to 12 weeks after third dose BNT162b2 (booster) vaccine. | 8-12 weeks after booster vaccine
Neutralizing geometric mean titers 8 to 12 weeks after third dose of BNT162b2 (booster) vaccine. | 8-12 weeks after booster vaccine

OTHER OUTCOMES:
The number of IFN-y-spot forming T cells SARS-CoV-2 specific after third dose of BNT162b2 (booster) vaccine. | 8-12 weeks after booster vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized IPD may be shared under institutional request if IRB requirements are met.

REFERENCES:
- [Derived] Dib M, Le Corre N, Ortiz C, Garcia D, Ferres M, Martinez-Valdebenito C, Ruiz-Tagle C, Ojeda MJ, Espinoza MA, Jara A, Arab JP, Rabagliati R, Vizcaya C, Ceballos ME, Sarmiento M, Mondaca S, Vinuela M, Pastore A, Szwarcfiter V, Galdames E, Barrera A, Castro P, Galvez NM, Soto JA, Bueno SM, Kalergis AM, Nervi B, Balcells ME. SARS-CoV-2 vaccine booster in solid organ transplant recipients previously immunised with inactivated versus mRNA vaccines: A prospective cohort study. Lancet Reg Health Am. 2022 Dec;16:100371. doi: 10.1016/j.lana.2022.100371. Epub 2022 Sep 23. PMID 36185969